CLINICAL TRIAL: NCT01223794
Title: Fall Risk Assessment for Inpatient
Status: Completed | Type: Observational
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Mei-Fen Taung, WanFang Hospital
Other Study IDs: 98101
Record Dates: First submitted 2010-10-17; First posted 2010-10-19 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2011-04

CONDITIONS: Accidental Falls
Keywords: Fall; all in surgical & Medical in-patient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Experimental Group: Fall in higher risk
- Control Group: Fall in lower risk

SUMMARY:
Goals and future prospects:

1. To finish the survey of the high risk factor ratios and high incidence rates associated with falls among inpatient fallers.
2. To investigate the risk factors associated with falls and the consequential analysis related to falls among inpatient fallers.
3. A good precautionary measure of falls will reduce damages and injuries for the fallers, especially inpatients welfare. Our accomplishments of this research proposal will provide sufficient information and reference for the precautionary strategies associated with fall incidents. More importantly, the experiences and results will be further explored and shared among all other hospitals.

DETAILED DESCRIPTION:
Introductions:

Fall is a very important and challenging question among acute care and long-term care facilities. The average incidence rate of fall is approximately 40% of total anomalous reports among hospitals in United States. Fallers may suffer many severe injuries, including fracture and brain concussions. Even fall had become interesting and popular topics for medical issues, the efforts of precaution for the fall incidents are still not evident. After Wanfang Hospital was established in 1997, the fall problems associated with inpatient fallers is one of most emphasizing issue in our medical cares. Since 1998, we began to implement policies in screening the risk factors associated with falls and to involve in the precautionary measures for the fallers. But the results come out not effectively.

Specific Aims:

The specific aims of this research proposal are the following:

1. Among inpatients, we will investigate the causes/reasons and risk factors associated with fallers and the incidence rates of falls. The consequences related to falls will also be studied.
2. We will evaluate our strategies on the efficacy of the precautionary measures for inpatients fallers.

Experimental design: The "Observational cohort experimental design" will be applied in this research proposal.

Data collections:

1. Data are collected mainly from wards of medicine and surgery. The project period is from 1/1/2009 to 12/31/2009.
2. The inpatients history, diagnosis, prescribed drugs, hemoglobin value, and blood sugar value of inpatients fallers will be collected and analyzed.
3. Associations between variables and falls among each individual faller will be assessed and evaluated thoroughly. If fall incident actually occurred, data on patient falls will be gathered within 48 hr and compared with each own relevant individual case by full evaluators.

Statistical analysis The Student-t test, Chi-square test, and one-way ANOVA will be preformed for the whole experimental data analysis.

Goals and future prospects:

1. To finish the survey of the high risk factor ratios and high incidence rates associated with falls among inpatient fallers.
2. To investigate the risk factors associated with falls and the consequential analysis related to falls among inpatient fallers.
3. A good precautionary measure of falls will reduce damages and injuries for the fallers, especially inpatients welfare. Our accomplishments of this research proposal will provide sufficient information and reference for the precautionary strategies associated with fall incidents. More importantly, the experiences and results will be further explored and shared among all other hospitals.

ELIGIBILITY:
Inclusion Criteria:

* above 18 years old
* Because in surgical department disease hospital
* The patient or the watcher may the country Taiwanese communication, consciousness clarity

Exclusion Criteria:

* Mental illness patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all in surgical & Medical in-patient
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2010-02; Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Fen Taung, Principal Investigator — Taipei Medical University WanFang Hospital
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan